CLINICAL TRIAL: NCT03826862
Title: Prospective Study on Image-guided Internal Iliac Vessels Dissection and Node-for-node for Selected Lateral Lymph Node Dissection in Middles-low Rectal Cancer
Brief Title: Lateral Lymph Node Dissection for Middle-low Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziqiang Wang,MD (Other)
Responsible Party: Sponsor-Investigator, Ziqiang Wang,MD, Clinical professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LLND-2018
Record Dates: First submitted 2019-01-25; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Rectal Cancer
Keywords: lateral lymph node dissection; node-by-node; rectal cancer; CT three-dimensional reconstruction; internal iliac vessels dissection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This group with intervention will be compared previous group without intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): All patients receive CT three-dimensional reconstruction before surgery.
  Interventions: Radiation: CT three-dimensional reconstruction
- control group (No Intervention): All patients did not receive CT three-dimensional before surgery

INTERVENTIONS:
Radiation: CT three-dimensional reconstruction — All patients will receive CT three dimensional reconstruction before surgery
  Arms: intervention group

SUMMARY:
The investigators will perform CT three-dimension reconstruction for middle-low rectal cancer patients who have enlarged lateral lymph nodes to recognize the variance of pelvic vessels, by which to help reduce operative time and blood loss, localize the lateral lymph nodes, improve the lymph node harvested and positive rate. Besides, The investigators will label the vessels near the interested node to achieve node-by-node for further investigation.

DETAILED DESCRIPTION:
CT three-dimensional reconstruction was performed for middle-low patients who had enlarged lateral lymph node before surgery. The main purpose is to recognize the track and variance of pelvic and iliac blood vessels. The investigators want to explore whether this method can help reduce operative time, unexpected injuries and blood loss, and The investigators also want to study whether it can help improve the lymph node harvested and positive rate during lateral lymph node dissection. Besides, The investigators want to perform node-by-node for enlarged lateral lymph node and CT three-dimensional reconstruction can help the investigators to localize and label the interested lymph node during operation. After node-by-node, The investigators can explore the accuracy of radiologists' and surgeons' judgement for lateral lymph node metastasis, and The investigators also want explore the best cut-off value of shorter diameter to predict lateral lymph node metastasis. Besides, The investigators want to perform texture analysis by combination radiology and pathology to find some useful parameters to predict lateral lymph node metastasis.

The investigators also want to explore the feasibility of dissecting the unilateral visceral branch of internal iliac vessels when performing lateral lymph node dissection.

The investigators will have a close follow-up for patients who have enlarged lateral lymph node but do not meet the criteria for lateral lymph node dissection. CT three-dimensional reconstruction can help The investigators recognize which parts' lateral lymph nodes have more potential possibility to metastasis and recurrence.

ELIGIBILITY:
Inclusion Criteria: 1) confirmed rectal cancer; 2) tumor located less than 10 cm from the anus verge; 3) have enlarged lateral lymph on preoperative CT/MRI

Exclusion Criteria: 1) patients who have severe liver or renal dysfunction;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
operative time | 2 year
  including total operative time and that for lateral lymph node
Blood loss | 2 year
  intraoperative blood loss
lateral lymph node harvested | 2 year
  lateral lymph node harvested
Accuracy of judgement for lateral lymph node metastasis | 2 year
  including radiologists' and surgeons' accuracy
Cut-off value of shorter diameter | 2 year
  The best cut-off value of shorter diameter for lateral lymph node dissection
vessels variances | October 1. 2018-December 31.2020
  The blood vessels variance of internal iliac vessels
postoperative complication | 2 year
  including urinary and sexual function

SECONDARY OUTCOMES:
local recurrence rate | 3 year
  local recurrence rate
overall survival | 3 year
  overall survival
disease-free survival | 3 year
  disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, MD, Study Chair — Department of Gastrointestinal Surgery, West China Hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided